CLINICAL TRIAL: NCT03469063
Title: Randomized Clinical Trial to Assess the Impact of AferBio® on Quality of Life and Toxicity to Chemotherapy in Patients With NSCLC Beginning Second-line Palliative Mono-chemotherapy
Brief Title: Impact of AferBio® on Quality of Life and Chemotherapy Toxicity in Lung Cancer Patients
Acronym: AFERBIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BarretosCH-20174
Record Dates: First submitted 2018-02-19; First posted 2018-03-19 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-02

CONDITIONS: Quality of Life; Infection; Drug Toxicity
MeSH Terms: conditions — Infections; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AferBio (Experimental): Daily oral AferBio (20 g/day, in sachets)
  Interventions: Dietary Supplement: AferBio
- Placebo (Placebo Comparator): Daily oral placebo (20 g/day, in sachets)
  Interventions: Dietary Supplement: AferBio

INTERVENTIONS:
Dietary Supplement: AferBio — Patients will use the product (AferBio/Placebo) once a day for seven days, and then twice a day, continuously (for a total of three months of use).

SUMMARY:
The AFERBIO study will evaluates safety and potential benefit of AferBio® in patients with non-small cell lung cancer undergoing at least a second-line palliative monochemotherapy. AferBio® is a fermented supplement in powder form obtained through biotechnological processes developed in Brazil. In this double-blind placebo-controlled randomized clinical trial, participants starting a new palliative regimen will be allocated to AferBio® or placebo. The primary aim will be to compare health-related QOL scores among the arms of the study over time.

ELIGIBILITY:
Inclusion Criteria:

* Age above or equal to 18 years, and below 75 years;
* Diagnosis of metastatic or recurrent NSCLC, beginning second-line palliative mono-chemotherapy treatment;
* Functional capacity (ECOG-PS) grade 0 - 2;
* Adequate hematological, kidney and liver function, as follows:

  * Total neutrophil count ≥ 1500/μL
  * Platelet count ≥ 100.000/μL
  * Hemoglobin ≥ 9 g/dL
  * Serum bilirubin ≤ 1.5 × upper limit of normal (ULN)
  * Patients with confirmed Gilbert's syndrome and serum bilirubin ≤ 3 × ULN
* Aspartate aminotransferase (AST), alanine transaminase (ALT), alkaline phosphatase ≤ 1.5 × ULN, serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min based on the Cockcroft-Gault equation:

  (140 - age) × (weight in Kkg) × (0.85) 72 × (serum creatinine in mg/dL)
* Absence of any emotional, family-related, sociological, or geographic condition that can potentially hamper adherence to the study protocol and the follow-up schedule;
* Capacity and willingness to adhere to the study visits and tests, and to adhere to the protocol, according to the researcher's evaluation.

Exclusion Criteria:

* Tube feeding, gastrostomy- or jejunostomy;
* Uncontrollable vomiting;
* Sexually active women of reproductive age, except for those who underwent surgical sterilization (e. g., tubal ligation);
* Intestinal obstruction or sub-obstruction;
* Known allergy to any of the components of the investigational product;
* Malabsorption syndrome or other condition that could interfere with enteric absorption;
* History of inflammation of the small or large intestine, previous or currently active (such as Crohn's disease or ulcerative colitis);
* Chronic diarrhea of any cause;
* Diagnosis of any chronic disease that, in the researcher's opinion, will interfere with the participation in the study;
* Known diagnosis of HIV -infection;
* Diagnosis of any chronic disease that changes the immune system and significantly increases the risk of infection;
* The need to use G-CSF already in the first chemotherapy cycle;
* Severe neuropsychiatric disease that prevents the patient from completing the study questionnaires, determined at the researcher's discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2018-06-28 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Health-related QOL scores over time. | Over time (during 90 days)
  To compare health-related QOL scores among the arms of the study over time.

SECONDARY OUTCOMES:
Toxicity | 3 months
  To compare the incidence of any given toxicity ≥ grade 3 (jointly and individually)
20% reduction in HRQOL | Along the study (3 months)
  To compare worsening-free survival of 20 % of the health-related QOL scores among the arms of the study;
Treatment delays | 3 months
  To compare the numbers of days of treatment delay due to toxicity, infections or worse performance status among the arms of the study;
Dose intensity | 3 months
  To compare the dose intensity (in mg/m2/week) among the arms of the study
Dose-reduction rates | 3 months
  To compare dose-reduction rates (≥ 20 %) and calculate dose reduction-free survival among the arms of the study;
Hospitalizations | 3 months
  To compare the number of hospitalizations among the arms of the study;
Infections | 3 months
  To compare the number of infections (any grade) among the arms of the study.
Use of anti-microbials | 3 months
  To compare the number of patients that used anti-microbials among the arms of the study.
Use of G-CSF | 3 months
  To compare the number of chemotherapy cycles with addition of granulocyte colony-stimulating factor (G-CSF) among the arms of the study.
Incidence of febrile neutropenia | 3 months
  To compare the incidence of febrile neutropenia among the arms of the study.
ECOG-PS worsening-free survival | Along the study (3 months)
  To compare worsening-free survival of the ECOG-PS (> 1 point) among the arms of the study
Nutritional status | Along the study (3 months)
  To compare nutritional status among the arms of the study
Antineoplastic response rates | 3 months
  To compare antineoplastic response rates among the arms of the study
Progression-free survival | 3 months
  To compare progression-free survival among the arms of the study
Adherence to AferBio® | 3 months
  To assess adherence to treatment with AferBio®

CONTACTS AND LOCATIONS:
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Almeida Preto D, Baston MT, Geraige CC, Augusto SB, de Oliveira MA, Mamere AE, Pinto GDJ, Dias JM, De Marchi PRM, Paiva BSR, Paiva CE. Impact of AferBio(R) on quality of life and chemotherapy toxicity in advanced lung cancer patients (AFERBIO study): protocol study for a phase II randomized controlled trial. BMC Cancer. 2019 Apr 25;19(1):382. doi: 10.1186/s12885-019-5599-z. PMID 31023257